CLINICAL TRIAL: NCT02906878
Title: Evaluation of the Effectiveness and Security of the Prophylactic Platelet Transfusion in Thrombocytopenic Patients Requiring the Placement of a Central Venous Catheter
Brief Title: Platelet Kinetics After Platelet Transfusion for the Placement of a Central Venous Catheter
Acronym: PLATCAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015-AO1924-45
Record Dates: First submitted 2016-07-05; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Thrombopenia; Central Venous Catheter Placement
Keywords: Intensive Care; Haematology; Platelets prophylactic transfusion
MeSH Terms: conditions — Thrombocytopenia | interventions — Platelet Transfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Platelets transfusion — Prophylactic platelet transfusion in thrombocytopenic patients for the placement of a central venous catheter

SUMMARY:
PLATCAT study's purpose is to evaluate platelet kinetics after platelet transfusion

ELIGIBILITY:
Inclusion Criteria:

* Admission en haematology unit
* Need for a central venous catheter
* Thrombopenia < 50 G/L

Exclusion Criteria:

* Patient protected by law
* Pregnant or breastfeeding women
* Peripheral thrombopenia
* Patient admitted in Intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haematology patients who needs a central venous catheter and with a non-auto immune thrombopenia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
72 hours thrombocythemia kinetics after a platelet transfusion | 72 hours post transfusion
  Blood drawing a H-1:00, H+0:10, H+1:00, H+4:00, H+24h00, H+72:00 Evaluation of platelets count on sodium citrate tube.

SECONDARY OUTCOMES:
Transfusion Safety - assessed by Troubles during process | One day after transfusion
  Troubles during process (pneumothorax, laying failure, hematoma) Hematoma at H+24:00 Immunisation anti HLA,HPA
Transfusion Efficacy | One month after transfusion
  Number of blood or platelets transfusion
Description of patients treatment | One week before and one month after transfusion
  Type of received chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEROLLE, MD PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No